CLINICAL TRIAL: NCT01460706
Title: PET/CT Imaging of Malignant Glioma With Somatostatin Analog 68Ga-DOTATOC
Brief Title: Imaging Malignant Glioma With 68Ga-DOTATOC PET/CT
Acronym: DOTAGLI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Heikki Minn, Chief Physician, Turku University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 77/180/2010
Record Dates: First submitted 2011-10-25; First posted 2011-10-27 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Glioma
Keywords: Glioma; 68Ga-DOTATOC; PET/CT; Somatostatin receptor
MeSH Terms: conditions — Glioma | interventions — Ga(III)-DOTATOC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 68Ga-DOTATOC (Experimental)
  Interventions: Drug: [68Ga]DOTATOC

INTERVENTIONS:
Drug: [68Ga]DOTATOC — 120MBq 68Ga-DOTATOC intravenously and PET/CT imaging. Performed once to a patient before the surgery.

SUMMARY:
The purpose of this study is to characterize tumour uptake of somatostatin analog 68Ga-DOTATOC in patients with either primary or recurrent malignant glioma. The investigators hypothesis is that some primary and recurrent malignant gliomas overexpress SST2 receptor which can be imaged with 68Ga-DOTATOC PET/CT. The investigators also hypothesize that tumor uptake of 68Ga-DOTATOC correlates with immunohistochemically determined SST2 receptor status of the tumor specimen.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 70 years old
* Language spoken: Finnish or Swedish
* Performance status: Karnofsky score 70 or better or WHO performance status 2 or better
* Supratentorial malignant glioma based on MRI imaging
* Supratentorial recurrent glioma based on MRI and/or [11C]methionine PET imaging
* Patients must be able to understand the meaning of the study and sign the appropriate Ethical Committee approved informed consent documents in the presence of the designated staff

Exclusion Criteria:

* Any medical or psychiatric condition that compromises the subject´s ability to participate in the study
* Any other significant disease including liver or renal disease
* Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Malignant glioma uptake of 68Ga-DOTATOC | within 90 minutes post-injection
  PET/CT imaging of the brain starts immediately after the intravenous bolus injection of 68Ga-DOTATOC. Dynamic PET/CT imaging is done over 60-min. A late 90-min scan will be obtained for selected patients. PET studies are analyzed by determining the Standardized Uptake Values (SUV) of the tumor using regions of interest (ROI) drawn both manually and automatically on the tumor.

SECONDARY OUTCOMES:
Immunohistochemical SST2 receptor status of the tumor specimen | After glioma surgery within 4 weeks of PET/CT imaging

CONTACTS AND LOCATIONS:
Overall Officials: Heikki RI Minn, M.D., Ph.D., Principal Investigator — Turku University Hospital
Locations (1):
- Turku PET Centre, Turku University Hospital, Turku, Finland

REFERENCES:
- [Derived] Kiviniemi A, Gardberg M, Frantzen J, Pesola M, Vuorinen V, Parkkola R, Tolvanen T, Suilamo S, Johansson J, Luoto P, Kemppainen J, Roivainen A, Minn H. Somatostatin receptor subtype 2 in high-grade gliomas: PET/CT with (68)Ga-DOTA-peptides, correlation to prognostic markers, and implications for targeted radiotherapy. EJNMMI Res. 2015 Apr 22;5:25. doi: 10.1186/s13550-015-0106-2. eCollection 2015. PMID 25977882